CLINICAL TRIAL: NCT01587820
Title: A Pilot/ Feasibility Study Comparing Response Rates of Intra-arterial and Intravenous Cisplatin Chemotherapy, Combined With Radiation, in Patients With Locally Advanced Carcinoma of the Oral Cavity and Oropharynx
Brief Title: Intra-arterial Versus Intravenous Cisplatin, Combined With Radiation, for Oral Cavity and Oropharynx Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROB-SCI 12-001
Record Dates: First submitted 2012-03-19; First posted 2012-04-30 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-07

CONDITIONS: Head and Neck Cancer
Keywords: cisplatin; RADPLAT; intra-arterial chemotherapy; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intra-arterial cisplatin and radiation (Experimental): 150 mg/m2 cisplatin given intra-arterially combined with sodium thiosulfate infusion given on days 1, 8, 15, for a total of 4 cycles, each cycle totaling 7 days and Radiotherapy: Primary tumor and upper neck will be treated with 2 Gy/fraction, once a day, five days a week to a total dose of 70 Gy/35 fractions/7 weeks
  Interventions: Drug: Intra-arterial cisplatin
- Intravenous cisplatin and radiation (Active Comparator): 100 mg/m2 cisplatin given intravenously once every 21 days (3 week cycle) for 3 cycles and Radiotherapy: Primary tumor and upper neck will be treated with 2 Gy/fraction, once a day, five days a week to a total dose of 70 Gy/35 fractions/7 weeks
  Interventions: Drug: Intravenous cisplatin

INTERVENTIONS:
Drug: Intra-arterial cisplatin — 150 mg/m2 cisplatin given intra-arterially combined with sodium thiosulfate infusion given on days 1, 8, 15, for a total of 4 cycles, each cycle totaling 7 days and Radiotherapy: Primary tumor and upper neck will be treated with 2 Gy/fraction, once a day, five days a week to a total dose of 70 Gy/35 fractions/7 weeks
  Arms: Intra-arterial cisplatin and radiation
Drug: Intravenous cisplatin — 100 mg/m2 cisplatin given intravenously once every 21 days (3 week cycle) for 3 cycles and Radiotherapy: Primary tumor and upper neck will be treated with 2 Gy/fraction, once a day, five days a week to a total dose of 70 Gy/35 fractions/7 weeks
  Arms: Intravenous cisplatin and radiation

SUMMARY:
This is a randomized, open-label investigator initiated pilot/ feasibility study comparing the effectiveness of intra-arterial administration of cisplatin therapy to intravenous administration of cisplatin when each is combined with the radiation therapy found in standard care. Participants will be randomized to either intra-arterial or intravenous cisplatin chemotherapy. This study is designed to determine whether a large scale study is practical in the investigators clinical setting. Approximately 10 subjects will be enrolled over a 2 year period.

DETAILED DESCRIPTION:
Head and neck malignancies represent a group of epithelial tumors that arise from the oral cavity, pharynx, and larynx and account for about 3 to 5% of all cancers in the United States. In 2010, an estimated 49,260 people (35,530 men and 13,730 women) will develop head and neck cancer, and an estimated 11,480 deaths (8,300 men and 3,180 women) will occur.

Three modalities of therapy have established roles in the treatment of carcinoma of the head and neck: chemotherapy, radiation therapy, and surgery. The choice of modality depends upon many factors such as the site and extent of the primary lesion, the likelihood of complete surgical resection, the presence of lymph node metastases, etc. Traditionally, smaller lesions (stage T1-T2) are effectively treated either, by surgical excision or irradiation whereas more advanced disease (T3-T4) is treated with combined surgery and radiation or chemoradiation. The goal of concurrent chemotherapy with radiation is to increase locoregional control and prevent distant metastases.

A specific concomitant chemoradiation protocol for head and neck cancer known as RADPLAT employs the pharmacologic principles and techniques described above. Capitalizing on the cisplatin-neutralizing agent sodium thiosulfate and its pharmacokinetic properties, enormous concentrations of cisplatin can be infused directly into large head and neck tumors through a targeted IA approach. In a Phase I study, it was determined that cisplatin could be safely administered to patients with advanced and recurrent head and neck cancer at a dose intensity of 150mg/m2/week.

The patient must be considered a clinical candidate for either intra-arterial or intravenous administration of cisplatin to be eligible for the study. Once enrolled and registered on the study, the subject will be randomized to either intravenous or intra-arterial administered cisplatin. Subjects will be assigned in a 1:1 ratio of intra-arterial versus intravenous administration. All patients will receive concurrent radiation therapy. Standard institutional practice will be applied for dose reduction and treatment of radiation therapy related toxicities.

A combination of lateral opposing fields will be used for the treatment of the primary tumor site and upper neck when three dimensional CRT is used and is not applicable for IMRT. A single anterior A-P field can be used to treat the lower neck below the primary tumor/upper neck. When there are positive nodes in the lower neck, an additional posterior field may be necessary to deliver a supplemental dose to the positive nodes. All fields must be treated on each treatment session.

The investigators will measure feasibility of the study protocol through enrollment and screen failure data. The study will test the hypothesis that intra-arterial cisplatin is more effective for patient outcomes in overall survival, disease free survival, cancer specific survival, rate of local and regional control of cancer, site of recurrence, organ preservation rate, toxicity, and correlative specimen availability.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Histologically or cytologically confirmed stage IV squamous cell carcinoma of the oral cavity or oropharynx staged according to AJCC guidelines
* T4 staged tumor with a tumor volume greater than or equal to 30 cc
* Nodal staging of N0 through 2a
* No evidence of distant metastatic disease, as determined by a negative PET scan or other clinically appropriate means
* Age ≥ 18
* Clinically eligible for both intra-arterial and intravenous administration of cisplatin
* Women of childbearing potential must have a negative pregnancy test.
* Agree to use adequate contraception prior to study entry and for the duration of study participation and for 3 months after study treatment ended
* Biopsiable via a transoral approach
* Life expectancy of at least 5 years
* ECOG performance status ≤ 2
* Measurable disease as defined by RECIST criteria
* Absolute neutrophil count ≥ 1,000/mm3
* Hemoglobin ≥ 8.0 g/dl
* Platelet count ≥ 100,000/mm3
* Leukocytes≥3500/mcL
* Total Bilirubin ≤ ULN of institution performing testing
* Creatinine within normal institutional limits

Exclusion Criteria:

* Radiologic evidence of bone destruction
* Tumor with involvement of cartilage or bone
* Requires bilateral IA infusion with radiologist determination that tumor extends across the midline in excess of 30% of the tumor volume
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents and pre-medications used in the study, including drugs formulated with polysorbate 80
* Allergy to cardiac catheterization contrast agents, in which antihistamines are not sufficient to suppress a reaction or severe enough to pose a significant danger to the subject
* History of stroke, CABG, or significant blockage of carotid arteries or coronary arteries or current blockage of coronary or carotid arteries equal to or in excess of 50% blockage; Interventional radiology must agree that the patient is a good candidate for catheterization.
* Intolerance to IV, IA, or radiation therapy treatment for any reason as determined by the procedural physician
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy
* Breast feeding women
* Prior or concurrent non-head and neck malignancies, excluding adequately treated basal or squamous cell cancer of the skin, in situ cervical cancer, stage I or II cancer from which the subject has been in complete remission for at least 12 months, any cancer from which the subject has been cancer free for 5 years
* Tumor site which cannot provide a biopsy in the clinic via punch or core needle biopsy performed
* Second primary head and neck tumor (concurrent or previous head and neck tumor unless it was a basal or squamous cell skin cancer)
* Unknown primary tumor site
* Prior surgery, chemotherapy, biologic or radiotherapy for a head or neck malignancy (excluding minor surgical procedures for skin cancer)
* History of surgery (non-oncologic) in the field of the tumor or treatment bed.
* Participation in an investigational treatment or intervention study within 90 days of screening visit
* calculated creatinine clearance less than 60 mL/min/1.73 m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
number of enrolled subjects | 2 years
  enrollment

SECONDARY OUTCOMES:
patient survival | 2 years
  patient survival data including overall survival, disease free survival, and cancer specific survival
rate of patient morbidity | 2 years
  rate of local and regional control of cancer, including site of recurrence and organ preservation rate

CONTACTS AND LOCATIONS:
Overall Officials: K. Thomas Robbins, MD, Principal Investigator — Southern Illinois University School of Medicine
Locations (2):
- United States (2):
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Simmons Cancer Institute at SIU School of Medicine, Springfield, Illinois

REFERENCES:
- [Background] Samant S, van den Brekel MW, Kies MS, Wan J, Robbins KT, Rosenthal DI, Rasch C, Weber RS. Concurrent chemoradiation for adenoid cystic carcinoma of the head and neck. Head Neck. 2012 Sep;34(9):1263-8. doi: 10.1002/hed.21905. Epub 2011 Nov 15. PMID 22083968
- [Background] Robbins KT, Howell SB, Williams JS. Intra-arterial chemotherapy for head and neck cancer: is there a verdict? Cancer. 2010 May 1;116(9):2068-70. doi: 10.1002/cncr.24930. No abstract available. PMID 20186833
- [Background] Robbins KT, Homma A. Intra-arterial chemotherapy for head and neck cancer: experiences from three continents. Surg Oncol Clin N Am. 2008 Oct;17(4):919-33, xi. doi: 10.1016/j.soc.2008.04.015. PMID 18722926
- [Background] Doweck I, Robbins KT, Samant S, Vieira F. Intra-arterial chemoradiation for T3-4 oral cavity cancer: treatment outcomes in comparison to oropharyngeal and hypopharyngeal carcinoma. World J Surg Oncol. 2008 Jan 14;6:2. doi: 10.1186/1477-7819-6-2. PMID 18194553
- [Background] Rabbani A, Hinerman RW, Schmalfuss IM, Amdur RJ, Morris CG, Peters KR, Robbins KT, Mendenhall WM. Radiotherapy and concomitant intraarterial cisplatin (RADPLAT) for advanced squamous cell carcinomas of the head and neck. Am J Clin Oncol. 2007 Jun;30(3):283-6. doi: 10.1097/01.coc.0000258118.38177.74. PMID 17551306
- See also: Simmons Cancer Institute at SIU School of Medicine — http://www.siumed.edu/cancer/